

# Statistical Analysis Plan (SAP) EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test

# AnteoTech LTD.

**Document reference number:** Version 1.0

Date: 23-Nov-2022



# **TABLE OF CONTENTS**

| 1. | SYN | IOPSIS OF STUDY DESIGN | 4 |
|----|-------|-----------------------------------------|---|
| | 1.1 | Purpose of Statistical Analysis Plan | 4 |
| | 1.2 | Clinical Performance Study Objectives | 4 |
| | 1.3 | Clinical Performance Study Design | 4 |
| | 1.4 | Endpoints | 4 |
| | 1.4. | 1 Primary endpoint | 4 |
| | 1.4.2 | 2 Secondary endpoint | 5 |
| 2. | ANA | ALYSIS CONSIDERATIONS | 6 |
| | 2.2 | Statistical Methods | 6 |
| | 2.3 | Endpoint Analysis | |
| | 2.3. | | |
| | 2.3.2 | 2 Secondary endpoint(s) | 7 |
| 3. | DES | SCRIPTIVE ENDPOINTS AND ADDITIONAL DATA | 9 |
| | 3.2 | Adverse Events | 9 |
| | 3.3 | Subject Early Termination | 9 |
| | 3.4 | Protocol Deviation | 9 |





| 5. | ACRONYMS AND ABBREVIATIONS | 11 |
|----|----------------------------------------|----|
| 4. | DOCUMENTATION AND OTHER CONSIDERATIONS | 10 |
| | 3.5 Number of Subject Imbalance | 9 |


Template CA-13.00.01-A




#### 1. SYNOPSIS OF STUDY DESIGN

#### 1.1 Purpose of Statistical Analysis Plan

This statistical analysis plan (SAP) is intended to provide a detailed and comprehensive description of the planned methodology and analysis to be used for the EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test Clinical Performance Study (CPS)

## 1.2 Clinical Performance Study Objectives

The objective of this CPS is to determine the diagnostic accuracy (sensitivity and specificity) of the EuGeni SARS-CoV-2 Antigen Rapid Diagnostic Test in the diagnosis of SARS-CoV-2 in specimens prospectively collected by healthcare professionals from subjects suspected of COVID-19 disease or with unknown COVID-19 status.

## 1.3 Clinical Performance Study Design

This CPS has been designed as a non-interventional, two-arm, prospective, non-randomized, open-label and multi-center study. Specimens can be prospectively collected by two different methods, which define the two arms of the study:

- 1. Nasopharyngeal specimen collection for comparison with gold-standard RT-PCR.
- 2. Combined nasal mid-turbinate and throat specimen collection for comparison with gold-standard RT-PCR.

| • |
|---|

#### 1.4 Endpoints

#### 1.4.1 Primary endpoint

The primary endpoint of this clinical performance study is to assess the EuGeni SARS-CoV-2 Ag RDT diagnostic accuracy, measured as the following:

| • | The diagnostic sensitivity of EuGeni SARS-CoV-2 Ag RDT, defined as the ability to identify the presence |
|---|---|
| | of a target marker associated with SARS-CoV-2, |
| | compared with gold-standard SARS-CoV-2 RT-PCR |






| • | The diagnostic specificity of EuGeni SARS-CoV-2 Ag RDT, defined as the ability to recognize the absence of a target marker associated with SARS CoV-2, compared with gold-standard SARS-CoV-2 RT- |
|---|---|
| | PCR. |
| 1.4.2 | Secondary endpoint |
| diagnos<br>and cor | condary endpoint of this clinical performance study is to compare the EuGeni SARS-CoV-2 Ag RDT stic accuracy (specificity and sensitivity) between the two specimen collection methods (nasopharyngeal mbined nasal mid-turbinate and throat) Randomization |
| 1.6 | Blinding |


Template CA-13.00.01-A

Page **5** of **18** 



#### 2. ANALYSIS CONSIDERATIONS

## 2.1 Analysis Populations

#### 2.1.1 Per-protocol (PP) population

| | | | population | includes | all | specimens | that | meet | the | study | eligibility | and | informed | consent |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| require | ements | | | | | | | | | | | | | ) |
| • | | | | | | | | | | | | | | |
| | ` | | | | | | | | | | | | | |
| 2.2 | Stat | istica | al Metho | ds | | | | | | | | | | |
| _ | _ | | | | | | | | | | | | | |

## 2.2.3 Survival analyses

Survival analyses do not apply to this CPS.

## 2.2.4 Regression

No regression analyses are planned for this CPS.

#### 2.3 Endpoint Analysis

#### 2.3.1 Primary endpoint(s)

The primary endpoint of this CPS evaluates the EuGeni SARS-CoV-2 Ag RDT diagnostic accuracy, which is defined in terms of sensitivity and specificity:

| The sensitivity is the ability to detect a target marker associated with SARS-CoV-2. The sensitivity means the capacity to detect positive samples from COVID-19 patients. |
|---|

• The specificity is the ability to recognize the absence of a target marker, associated with SARS-CoV-2, which means the capacity to detect true negative samples of COVID-19.

Template CA-13.00.01-A 






Template CA-13.00.01-A




| _ | |
|---|---|
| 2.7 | Timing of Analysis |
| | tion to the interim analysis described above, the study endpoints will be assessed after all specimens are sed and analyzed by both the investigational device and the gold-standard RT-PCR technique, |
| 2.9 | Subgroups of Analysis |
| Subgro | oup analyses in the context of this CPS will be performed |
| differen | according to a specimen characteristics, which may include: |
| - | The viral load, determined by the Ct value obtained in the RT-PCR analysis. |
| - | Days from symptom onset. |
| - | |
| ĕ | |

# 2.14 Exploratory Analysis

No exploratory analyses are considered in this CPS.

Template CA-13.00.01-A 



# 3. DESCRIPTIVE ENDPOINTS AND ADDITIONAL DATA

| 3.2 Adverse Events |
|---|
| All the AEs, SAEs, adverse device effects (ADEs), serious adverse device effects (SADEs), unanticipated adverse device effects (UADEs), and unanticipated serious adverse device effects (USADEs) will be summarized for all subjects who are enrolled in this CPS |
| 3.3 Subject Early Termination |
| There is no formal statistical rule defined for early termination of the CPS for insufficient performance of the tested device. |
| 3.4 Protocol Deviation |
| Protocol deviations will be summarized by major and minor categories for subjects in whom a protocol deviation was reported. |
| 3.5 Number of Subject Imbalance |
| All efforts will be made to maintain a balanced enrollment among the participating sites. |


Template CA-13.00.01-A







# 5. ACRONYMS AND ABBREVIATIONS

| Acronym or Abbreviation | Complete Phrase or Definition |
|-------------------------|---------------------------------------------------|
| AE | Adverse Event |
| CPS | Clinical Performance Study |
| CPSP | Clinical Performance Study Protocol |
| FN | False Negative |
| FP | False Positive |
| RAT | Rapid Antigen Test |
| RT-PCR | Reverse Transcription - Polymerase Chain Reaction |
| TN | True Negative |
| TP | True Positive |
| SAE | Serious Adverse Event |
| SAP | Statical Analysis Plan |


Template CA-13.00.01-A






| · |
|---|




Template CA-13.00.01-A




| • |
|---|
| • |
| • |
| • |


Template CA-13.00.01-A







| 1 | l |
|---|---|


Template CA-13.00.01-A

Page **16** of **18** 



| l |
|---|


Template CA-13.00.01-A




